CLINICAL TRIAL: NCT05155319
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Dose-Escalation Study Evaluating Safety and Immunogenicity of Influenza A Hemagglutinin Stabilized Stem Nanoparticle Vaccine Candidate in Healthy Adults
Brief Title: Universal Influenza A Vaccine in Healthy Adults
Acronym: EBS-UFV-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EBS-UFV-001
Record Dates: First submitted 2021-11-25; First posted 2021-12-13 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Human Influenza
Keywords: universal; universal influenza vaccine; phase 1; randomized; double-blind; placebo
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1, 1A (Active Comparator): Low dose (Day 1) plus placebo (Day 22)
  Interventions: Biological: UFluA 20 µg each antigen/dose; Biological: Placebo
- Cohort 1, 1B (Active Comparator): Low dose (Day 1) plus low dose (Day 22)
  Interventions: Biological: UFluA 20 µg each antigen/dose
- Cohort 1, 1C (Placebo Comparator): Placebo (Day 1) plus Placebo (Day 22)
  Interventions: Biological: Placebo
- Cohort 2, 2A (Active Comparator): High dose (Day 1) plus placebo (Day 22)
  Interventions: Biological: UFluA 60 µg each antigen/dose; Biological: Placebo
- Cohort 2, 2B (Active Comparator): High dose (Day 1) plus high dose (Day 22)
  Interventions: Biological: UFluA 60 µg each antigen/dose
- Cohort 2, 2C (Placebo Comparator): Placebo (Day 1) plus Placebo (Day 22)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: UFluA 20 µg each antigen/dose — Low dose
  Arms: Cohort 1, 1A; Cohort 1, 1B
Biological: UFluA 60 µg each antigen/dose — High Dose
  Arms: Cohort 2, 2A; Cohort 2, 2B
Biological: Placebo — Placebo
  Arms: Cohort 1, 1A; Cohort 1, 1C; Cohort 2, 2A; Cohort 2, 2C

SUMMARY:
The goal of this Phase 1, single- center, randomized, double blind, placebo-controlled dose-escalation study is to evaluate the safety, tolerability and immunogenicity of UFluA vaccine candidate at two dose levels and two schedules in healthy adult (18-45-year-old, inclusive) male and non-pregnant female subjects.

DETAILED DESCRIPTION:
A total of 60 healthy adult subjects will be enrolled in the study and followed through Day 337 (i.e., up to 48 weeks after first dose). Subjects will be enrolled into two study cohorts to receive either a low dose (Cohort 1; n=30 receives) or high dose (Cohort 2; n=30) of adjuvanted UFluA or placebo (saline), administered intramuscularly (IM) as single dose or as two doses (administered 21 days apart).

UFluA is comprised of DP-UFluA (1:1 A1-ssnp and A2-ssnp antigens) and contains aluminum hydroxide and CpG adjuvants.

Primary Objective:

To evaluate safety and tolerability of UFluA IM administration in healthy adults.

Secondary Objectives:

To assess anti-hemagglutinin humoral immune responses in healthy adults who receive UFluA. To assess ferritin (Helicobacter pylori and human) immune response in healthy adults who receive UFluA.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults (18-45 years of age, inclusive) at the Screening visit.
* Body mass index of 18.5-32.0 kg/m^2 (inclusive) at the Screening visit.
* Healthy, based on medical history (no chronic disease, no chronic therapy, no ongoing acute condition within four weeks prior to dosing as per PI [or designee] discretion), normal PE (no clinically significant findings in the opinion of the PI [or designee]), no clinically significant findings on screening electrocardiogram (ECG) and laboratory assessments in the opinion of the PI [or designee].
* Females must not be pregnant or trying to become pregnant.
* Both male and female subjects agree to acceptable forms of birth control. Male subjects must not donate sperm for the duration of the study.

Exclusion Criteria:

* Enrollment in an interventional study and/or receipt of any investigational product within 30 days prior to screening visit or during the study.
* Currently breastfeeding or planning to be breastfeeding during the study.
* History of severe allergic reaction(s) or anaphylaxis.
* Known allergy to any component of the vaccine.
* History of any known immunodeficiency or immunocompromising condition that could impact response to administration of the investigational product (e.g., leukemia, lymphoma, malignancy, renal failure, asplenia, diabetes mellitus, alcoholic cirrhosis).
* Receipt or anticipated receipt of blood products from 180 days prior to the Screening visit through 90 days following administration of IP.
* Positive laboratory evidence of current infection at the Screening visit with HIV 1 and 2 (as determined by HIV 1/2 antibody test), HCV (as determined by HCV antibody test), or HBV [as determined by HBV surface antigen (HBsAg) test]. Note: positive anti-HCV antibody result along with a negative HCV PCR result would not be exclusionary.
* Any clinically significant abnormalities in rhythm, conduction, or morphology of the resting 12-lead electrocardiogram (ECG) based on the PI's (or designee's) review of tracing results at the Screening visit. [Non-pathologic sinus bradycardia (heart rate must be >40 beats per minute) is allowed].
* Receipt or anticipated receipt of the seasonal influenza vaccination from up to 90 days prior to dosing and through up to 30 days following the last dose administration.
* Receipt or anticipated receipt of any COVID-19 vaccine from up to 14 days prior to dosing and through up to 30 days following the last dose administration.
* Receipt or anticipated receipt of any other vaccines from up to 90 days prior to dosing and through up to 30 days following last dose administration of investigational product.
* Receipt or anticipated receipt of systemic immunomodulatory agents or other immune modifying drugs (including systemic corticosteroids exceeding 20 mg/day for ≥14 days) and antineoplastic agents from up to six months prior to dosing and through the entire duration of the study.
* Planned medical procedure(s) that will impact study compliance during the follow-up period.
* Positive urine drug screen test or any evidence of ongoing drug abuse or dependence (including alcohol), or recent history over the past five years of treatment for alcohol or drug abuse.
* Planning to donate bone marrow, blood, and blood products from the time of screening until 3 months after receiving the last dose.
* Have a tattoo/scar/birthmark or any other skin condition affecting the deltoid area that may interfere with injection site assessments.
* History of H. pylori infection or documented iron deficiency within the past five years.
* An opinion of the PI (or designee) that it would not be in the best interest of the subject to allow participation in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Safety of the UFluA vaccine following one of four dose schedules as evaluated through adverse events (AEs), serious adverse events (SAEs), adverse events of special interest (AESIs) and medically attended adverse events (MAAEs). | 48 weeks
  Incidence of AEs up to 4 weeks after last dose. Incidence of SAEs up to 48 weeks of study follow-up. Incidence of AESIs up to 48 weeks of study follow-up. Incidence of MAAEs up to 48 weeks of study follow-up.
Local and systemic reactogenicity of UFluA vaccination following one of four dose schedules. | seven days after each vaccination
  Incidences of local reactogenicity events up to 7 days after each vaccination. Incidences of systemic reactogenicity events up to 7 days after each vaccination.

SECONDARY OUTCOMES:
Anti-H. pylori ferritin immune response to UFluA vaccination. | up to 4 weeks after the last vaccination.
  Anti-H-pylori ferritin antibody titers at multiple timepoints up to 4 weeks after the last vaccination.
Anti-human ferritin immune response to UFluA vaccination. | up to 4 weeks after the last vaccination.
  Anti-human ferritin antibody levels at multiple timepoints up to 4 weeks after the last vaccination.
Humoral immune response to A1 influenza antigen following UFluA vaccination. | up to 4 weeks after the last vaccination.
  Peak anti-A1 stem binding antibody titers (as measured by an immunoassay) at multiple timepoints up to 4 weeks after the last vaccination.
Humoral immune response to A2 influenza antigen following UFluA vaccination. | up to 4 weeks after the last vaccination.
  Peak anti-A2 stem binding antibody titers (as measured by an immunoassay) at multiple timepoints up to 4 weeks after the last vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: James McCarthy, MD, Study Director — Emergent BioSolutions
Locations (2):
- Australia (2):
  - Northern Beaches Clinical Research, Brookvale, New South Wales
  - Linear Clinical Research, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No